CLINICAL TRIAL: NCT04268199
Title: A Multicentre, Non-Blinded Study Exploring Self-Administration of Chemotherapy in the Home Environment
Acronym: EASE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EASE
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Myeloma; Myeloma Multiple
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self Injection of Bortezomib (Other): Subcutaneous self administration of bortezomib
  Interventions: Drug: Bortezomib Injection

INTERVENTIONS:
Drug: Bortezomib Injection — Subcutaneous injection
  Other Names: Velcade

SUMMARY:
This study is to see if the standard of care subcutaneous injection of bortezomib can safely be administered at home by the patient or caregiver. All tests and assessments are based on standard of care procedures.

DETAILED DESCRIPTION:
Chemotherapy for malignancies is predominantly prescribed and delivered in a tertiary hospital and/or cancer centre setting. However, with modern chemotherapy, with a reduced side effect profile, this paradigm should be challenged. Indeed, the use of methotrexate and other biologics (a form of chemotherapy) in the Rheumatologic setting is commonly delivered effectively and safely in the community.

Taken together, a hospital-based model of chemotherapy delivery may not be warranted in all circumstances. Moreover, the use of this current model invariably discounts the time commitments, needs of patients and caregivers, as well as while not addressing the emerging concerns regarding system capacity, efficiency and effectiveness of safe chemotherapy delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged 18 years old or older with a diagnosis of symptomatic myeloma,
* Stable clinical status as deemed by responsible investigator,
* Personally (or caregiver) willing and deemed capable to self-administer with teaching,
* Previously received more than 4 injections of bortezomib within the hospital and/or cancer centre environment,
* Signed informed consent.

Exclusion Criteria:

* Currently participating in clinical trials that includes the use of bortezomib,
* History of allergic reactions to bortezomib,
* History of bleeding attributable to bortezomib,
* History of greater than or equal to grade 3 side effects attributable to bortezomib,
* Clinically deemed unlikely to be compliant with therapy by responsible investigator,
* Life expectancy anticipated to be less than 6 months,
* Deemed geographically inaccessible to receive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients able to self-administer | 2 years from study start
  Number of eligible patients availing of self-administration
Myeloma response outcomes | 2 years from study start
  Myeloma outcomes as per International Myeloma Foundation Response (IMWG) Criteria. For the purposes of this trial, best response will be documented.
Adverse events great than grade 3 | 2 years from study start
  Adverse event documentation as per CTCAE version 5.0 scales of greater than grade 3
Number of patients with missed doses | 2 years from study start
  Proportion of missed doses
Patient Satisfaction and Quality of Life Survey 1 | 2 years from study start
  Patient Satisfaction Surveys - FACIT-TS-PS (Functional Assessment of Chronic Illness Therapy)
Patient Satisfaction and Quality of Life Survey 2 | 2 years from study start
  Patient Satisfaction Surveys - CQOLC (Caregiver Quality of Life - Cancer)
Patient Satisfaction and Quality of Life Survey 3 | 2 years from study start
  Patient Satisfaction Surveys - EORTC QLQ-MY20 (European Organization of Research and Treatment of Cancer - Quality of Life)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tay, MD, Principal Investigator — Arthur J.E. Child Comprehensive Cancer Centre
Locations (2):
- Canada (2):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No